CLINICAL TRIAL: NCT05739084
Title: [RADIOSARC] Searching for Specific Gene Signature(s) of Sensitivity/Resistance to Neoadjuvant Radiotherapy in Adults Patients With Resectable Soft Tissue Sarcomas of Limbs
Brief Title: Gene Signatures Searching of Sensitivity/Resistance to Neoadjuvant Radiotherapy in Patients With Resectable STS
Acronym: RADIOSARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET21-240 [RADIOSARC]; GDPR registration Number (Other: R201-004-171)
Record Dates: First submitted 2023-01-26; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Soft Tissue Sarcomas
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Available FFPE Tumour samples at diagnosis and surgery from respectively Retrospective cohort [200 patients] and Propective Cohort [100 patients]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: A total sample size of 200 patients is expected in the retrospective thanks to the NETSARC/ CONTICABASE databases (French sarcoma reference network)
  Interventions: Radiation: pre-operative radiation; Procedure: Standard surgery after rpreoprative radiation
- Prospective cohort: To ensure an external validation, patients from NETsarc centers experiencing preoperative RT will be prospectively accrued and transcriptomic signature will be tested.
  Up to 100 patients will be enrolled in this prospective cohort.
  Interventions: Radiation: pre-operative radiation; Procedure: Standard surgery after rpreoprative radiation

INTERVENTIONS:
Radiation: pre-operative radiation — As per standard of care and institutional guidelines
Procedure: Standard surgery after rpreoprative radiation — As per standard of care and institutional guidelines

SUMMARY:
To date, the radiation oncologist are missing biomarkers predictive of response/resistance to RT in order to identify patients who may benefit from RT and personalize the RT schedule. Our proposal is to conduct a cohort study aiming at identifying transcriptomic biomarkers predictive of sensitivity and/or resistance to RT in limbs STS patients

DETAILED DESCRIPTION:
Whether RT should be performed pre or post-operatively is still a debated question. To date, the radiation oncologist are missing signature of response/resistance to RT in order to identify patients who may benefit from RT and personalize the RT schedule. Therefore, predicting the likelihood of response/resistance to RT is essential. The individual exploration with high-throughput approaches will participate in describing biological mechanisms involved in STS tumor cell pan-resistance, thus identifying potential molecular targets that could be inhibited to reverse intrinsic radioresistance. In this context, our proposal is to conduct a cohort study aiming at identifying transcriptomic signature predictive of sensitivity and/or resistance to RT in limbs STS patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years at time of non-opposition to participate to the study
* Patient with documented non-opposition to participate to the study.
* Patient with histologically and cytologically confirmed diagnosis with STS (..)
* Patient with availability of FFPE tumor block from initial diagnosis biopsy (mandatory) and surgery specimen (optional).
* Patients with tumor FFPE samples prepared with the last 4 years
* Patient with evaluable tumor sample meeting the following quality/quantity control criteria (..)

Exclusion Criteria:

* Patients with metastatic soft tissue sarcoma at diagnosis
* Patients with exclusive radiotherapy without surgical resection
* Patients receiving neo adjuvant systemic treatment (chemotherapy, immunotherapy, targeted therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Soft tissus sarcoma who underwent/undergo to preoperative Radiation and for whom resected tumour specimen is available.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-11-23 (Estimated)

PRIMARY OUTCOMES:
To define a transcriptomic signature of histological response to radiotherapy in STS patients using the percentage of residual viable cells as a clinical meaningful endpoint | 36 months
  Gene expression signature using RNAseq correlated to the percentage of residual viable cells on surgery specimen to define histological response.

SECONDARY OUTCOMES:
To identify biomarkers of sensitivity or resistance to radiotherapy in STS patients using additional clinical endpoints | 36 months
  Gene expression signature using RNAseq correlated to the percentage of necrosis, the percentage of fibrosis, the local control at 1 and 2 years (1- and 2-year local / distant recurrence-free survival, the time To Relapse (TTR), the Disease Free Survival (DFS), The Quality of resection level based on the residual tumor (R) classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No